CLINICAL TRIAL: NCT01316289
Title: Quality of Fracture Reduction and Its Influence on Functional Outcome in Patients With Pilon Fractures - a Prospective Multicenter Case Series
Brief Title: Pilon Fracture Reduction and Functional Outcome
Status: Completed | Type: Observational
Sponsor: AO Clinical Investigation and Publishing Documentation (Other)
Responsible Party: Sponsor
Organization: AO Innovation Translation Center (Other)
Other Study IDs: Pilon
Record Dates: First submitted 2011-03-14; First posted 2011-03-16 (Estimated); Last update posted 2020-08-13 (Actual); Status verified 2018-01

CONDITIONS: Pilon Fracture of Tibia
Keywords: tibial fractures; pilon; pilon fractures; tibial plafond; reduction quality; anatomical reduction; functional outcome; ankle joint
MeSH Terms: conditions — Tibial Fractures

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This prospective case series will essentially examine the influence of reduction quality on the primary functional outcome (as assessed using the FAAM) of patients with pilon fractures treated with plate fixation.

The plates used in this trial can be chosen according to the preferences of the surgeon.

DETAILED DESCRIPTION:
A prospective case series to examine the influence of reduction quality on the primary functional outcome (as assessed using the FAAM) of patients with pilon fractures treated with plate fixation. Radiological parameters including single/combined alignment and various articular measurements will also be validated according to their reliability. The sensitivity of the effects of reduction quality on functional outcome, and an extended evaluation of patient-rated functional and social outcomes as well as their outcome expectations will also be assessed as part of the secondary study aims.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years and older
* Patients with a unilateral intraarticular pilon fracture of the distal tibia classified according to AO: AO 43 - B1, B2 and B3 (partial intraarticular) AO 43 - C1, C2 and C3 (total intraarticular)
* Definitive fracture fixation with a plate within 4 weeks after accident (Temporary fixation with an external fixator, cast or traction is allowed)
* Signed written informed consent (by the patients) and agreement to attend the planned FU evaluations

Exclusion Criteria:

* Contralateral fracture of the distal half of the tibia/fibula/talus
* Pathologic fracture
* Severe Polytrauma: Injury Severity Score (ISS) > 28
* Preexisting severe vascular disease (chronic venous insufficiency, chronic arterial occlusive disease)
* Drug or alcohol abuse
* American Society of Anesthesiologists (ASA) class V and VI
* Inability to walk independently prior to injury event
* Neurological and psychiatric disorders that would preclude reliable assessment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with pilon fractures that fulfill the following inclusion and exclusion criteria
Sampling Method: Probability Sample
Enrollment: 117 (Actual)
Dates: Start 2011-11 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Examine the influence of reduction quality on the primary functional outcome (as assessed using the Foot and Ankle Ability Measure (FAAM)) of patients with pilon fractures treated with plate fixation. | 2 years
  The most important predictors of functional outcome after pilon fracture will be identified by evaluating the influence of radiologically assessed parameters of reduction quality and other factors (age, high/low energy trauma, AO fracture type, open/closed fracture, delay between trauma and definitive fracture fixation) on the FAAM. In parallel, the radiological parameters will also be validated with respect to their reliability.

SECONDARY OUTCOMES:
Surgical details | 1 year
  * Length of surgery (skin-to-skin time)
  * Type of implant used
  * Use of bone graft
  * Soft tissue or wound-related procedures (eg, debridement, free flap, local flap, split skin graft)
Pre- and postoperative treatment | 1 year
  Perioperative management data will include documentation of the use of thromboprophylaxis or prophylactic antibiotics, therapeutic antibiotics and pain medication including nonsteroidal antiinflammatory drugs (NSAID).
To assess whether patient and surgeon expectations are met with regard to the trauma outcome | 1 year
  Trauma expectations factor (TEF) to assess the patient and surgeon expectations about the outcome of the treatment

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Sommer, MD, Principal Investigator — Cantonal Hospital Graubuenden; Martin Schuler, PhD, Study Director — AO Clinical Investigation and Documentation, Davos, Switzerland
Locations (9):
- United States (4):
  - Indiana Orthopaedic Hospital, Indianapolis, Indiana
  - University of Minnesota, Saint Paul, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Harborview Medical Center, Seattle, Washington
- Medical University Innsbruck, Innsbruck, Austria
- Universidade de São Paulo - Faculdade de Medicina, São Paulo, CEP, Brazil
- Switzerland (3):
  - Cantonal Hospital Graubuenden, Chur
  - Cantonal Hospital Luzern, Lucerne
  - Cantonal Hospital Winterthur, Winterthur